CLINICAL TRIAL: NCT06764173
Title: The Difference in Health Outcomes After Drinking Cow's Milk Compared to Oat Milk - a Pilot Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Institute of Marine Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 712892
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-06

CONDITIONS: Plant-based Milk; Iodine Nutrition Status; Lipids
Keywords: Iodine nutrition status; Blood lipids; oat milk
MeSH Terms: interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cow's milk (Active Comparator): 6 dl of cow's milk daily
  Interventions: Other: Oat drink; Other: Cow's milk
- Oat drink (Experimental): 6 dl of Oat drink daily
  Interventions: Other: Oat drink; Other: Cow's milk

INTERVENTIONS:
Other: Oat drink — 6 dl of oat drink daily
Other: Cow's milk — 6 dl of cow's milk daily

SUMMARY:
A new dietary trend is switching from cow's milk to plant-based milk alternatives, driven by the belief that this switch is beneficial for health reasons in addition to the sustainability aspect of a plant-based diet. The trend of using plant-based milk alternatives is especially popular among young women, of whom iodine nutrition also is of concern, both globally and in Norway. Some of the plant-based alternatives are fortified with iodine, but both the bio-availability and whether is feasible to consume large enough amounts of the milk to provide an adequate iodine intake is unknown. Another aspect is that the effect of cow's milk intake on blood lipids has been widely studied, however, there is a lack of studies on the effect of oat milk consumption on blood lipids.

DETAILED DESCRIPTION:
The aim of this study is two-fold

1. To compare the iodine nutrition in those drinking cow's milk compared to oat milk
2. To compare the levels of blood lipids in those drinking cow's milk compared to oat milk

Recruitment Women aged 18-40 years deemed eligible according to the inclusion and exclusion criteria will be asked to participate in the study. The recruitment will occur at the University of Bergen during the fall of 2024. Those willing to participate will contact the study personal by a digital form. Before participation, signed informed consent must be provided.

Participants who uses dietary supplements will be asked to cease these during the intervention. The exception is those with clinical deficiency e.g. anemia.

Sample size This is a pilot study testing both the feasibility of the interventions and if we observe any changes in the outcomes. To our knowledge, no trials have been conducted comparing cow's milk and oat milk before. Hypothesizing that oat milk will decrease total cholesterol due to its content of beta-glucans and a higher content of PUFAS compared to cow's milk. For the cow's milk group, we expect the total cholesterol in the cow's milk group to stay the same before and after intervention. A mean difference of 0.6 mmol/l between the groups, will need groups of 174 with an alpha of 0.05 and power of 80%. Due to the limitations and time frame of a master thesis, we propose 15 persons per arm, thus including 30-40 participants. In our experience with similar intervention studies in the same group of participants, this sample size is feasible within the timeframe of a master's thesis.

Study design A pilot randomized study design will be performed, where the participants will be randomly divided into groups to either drink cow's milk or oat milk for 4 weeks in a dose of 6 dl per day, which corresponds to the dietary recommendation of "three portions of dairy products a day". The cow milk and oat milk will be provided to the participants and handed out in regular time intervals from the study center. The participants should not make any other changes to their habitual diet. Blood and urine samples will be collected at the Research Unit for Health Surveys. Additionally, the performance of a wearable patch for hydration monitoring (https://www.modesensors.com/) will be assessed in a subsample of 8 participants.

Measurements Anthropometric measurements Body weight and height will be measured at baseline, and body weight again at the end visit.

Dietary assessment 24-hour recalls will be performed several times during the intervention period to assess compliance with the intervention, monitor any deviations from habitual dietary intake, and to be able to calculate iodine intake from the diet.

Iodine nutrition 24-hour urine will be collected at baseline and after two weeks of intervention. In addition, two spot urine samples will be collected at baseline. The urine samples will be analyzed for iodine concentration (UIC) with ICP-MS at the Institute of Marine Research. In addition, creatinine and osmolarity will be measured both in the spot and 24-hour urine samples. Both thyroglobulin, TSH, fT3, and fT4 will be measured in serum at baseline and end visit. Iodine intake from the diet will be calculated based on the repeated 24-hour recalls. The participants are asked to keep a record of every bathroom visit and if there are any deviations (e.g. spillage).

Blood lipids Both triacylglycerol, total cholesterol, LDL, and HDL cholesterol will be measured at baseline and the end visit. All blood samples will be analyzed at the MBF at Haukeland University Hospital.

Compliance To assess compliance with the intervention milk, the participant is asked to fill in a compliance journal of their daily intake.

Ethics and safety Participants are provided with information about the study both orally and in writing and must sign a consent form to be included in the study before the baseline visit. The principle of the Declaration of Helsinki will be applied. The participants can withdraw from the study at any time without explanation.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-40 years
* healthy
* habitual milk drinkers

Exclusion Criteria:

* pregnant or lactating
* known thyroid disease
* planning to conceive

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Iodine nutrition | Basline and end of intervention after 4 weeks
  24-hr urine collection, 2 x spot urine, TSH, fT4, fT3, dietary iodine intake by 24-hour recall interview
Blood lipids | Basline and end of intervention after 4 weeks
  s-HDL, s-LDL, s-total cholesterol, s-triacylglyserol

SECONDARY OUTCOMES:
Body weight | Basline and end of intervention after 4 weeks
  Weight change during the study period
Hydration status | Basline and end of intervention after 4 weeks
  A sub-group of particiants will have their hydration status measure by a hydration sensor, osmolarity in the 24-hour urine, spot urine samples, electrolytes measure in blood

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Rosendahl-Riise, PhD, Principal Investigator — University of Bergen
Locations (1):
- Research Unit for Health Surveys, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
This is a pilot study with limited number of participants.